CLINICAL TRIAL: NCT06728384
Title: Remodeling of Distal Coronary Vessel in Chronic Total Occlusions: Prediction Based on Hemodynamic Coronary Parameters
Acronym: CTO-VR
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 111578
Record Dates: First submitted 2024-12-06; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Chronic Total Occlusion (CTO); Percutaneous Coronary Intervention (PCI); Fractional Flow Reserve; Quantitative Coronary Analysis; Absolute Flow Measurement; Optical Coherence Tomography (OCT)
Keywords: Chronic Total Occlusion; Percutaneous Coronary Intervention; Quantitative coronary analysis; Absolute flow measurement; Optical Coherence Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- CTO patients undergoing FFR collateral, Absolute flow and OCT measurements: FFR collateral will be measured by measuring the wedge pressure distal from the occlusion, and after stent implantation by creating a balloon-over-the-wire occlusion.
  MLD will be measured with quantitative coronary analysis (QCA)
  Absolute flow will be measured by using a rayflow catheter with a pressure wire, and by using the Coroventis system.
  OCT will be performed during follow-up, using an OCT catheter and perform a pullback through the entire stent trajectory.

SUMMARY:
Background Revascularization of a chronic total occlusion (CTO) has gained popularity last decade. After recanalization there is an acute gain in vessel diameter, as well as a late lumen gain distal to the stent as a result of positive remodeling. The evolution of a recanalized CTO-vessel is however diverse. Several studies are performed to measure distal lumen gain and hemodynamic coronary parameters of a recanalized CTO, including the novel measurement Absolute Flow. Although the results seem promising, an association between those parameters and distal vessel lumen gain has never been found. The aim of this study is to understand the remodeling of the distal coronary vessel in relation with hemodynamic coronary parameters, establishing baseline predictive factors, adding new information about coronary physiology.

Objectives:

To establish baseline predictive factors for acute and late lumen growth after successful opening of chronic total occlusions. Secondary objectives are 1) Identifying the relation between change in absolute microvascular resistance and late change distal lumen diameter at the end of the index procedure and at 3 months follow-up, 2) Identifying the relation between late lumen growth and stent malapposition, assessed using Optical Coherence Tomography (OCT) and 3) Identifying the relation between angina-related symptoms, assessed using the Seattle Angina Questionnaire-7 (SAQ-7), and absolute microvascular resistance.

Hypothesis:

Acute and late lumen growth are dependent on preprocedural distal coronary artery perfusion pressure, decrease in microvascular resistance and growth of absolute antegrade flow. Late lumen growth predisposes for late stent malapposition.

Study design:

A single-center, prospective, observational cohort study. The center performing this study will be the Radboudumc.

Study Population:

30 patients scheduled for an elective revascularization procedure of a CTO and Heart-team consensus for the indication of a CTO treatment.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled elective revascularization procedure of a CTO, defined as a complete obstruction of a coronary artery with TIMI-0 or TIMI-1 flow and occlusion duration of at least 3 months
* Heart-team consensus for the indication of a CTO treatment, based on viability and ischemia testing (using TTE or MRI)
* Able to give valid, written informed consent

Exclusion Criteria:

* Unsuccessful crossing of the lesion during PCI
* Renal insufficiency defined as eGFR < 30 ml/min
* Contra-indications to intravenous adenosine
* < 18 years of age
* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 30 patients scheduled for an elective revascularization procedure of a CTO and Heart-team consensus for the indication of a CTO treatment
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-08-28 (Actual)

PRIMARY OUTCOMES:
Acute FFR collateral change | 30 minutes
  Changes in collateral function in rest and hyperaemic state, measured before recanalization and after recanalization
Late FFR collateral change | 3 months
  Changes in collateral function in rest and hyperaemic state, measured after recanalization and at 3 months follow-up
Acute MLD change | 30 minutes
  Changes in mean lumen diameter of the treated vessel, measured up to 5 mm distal to the occlusion before recanalization and distal to the stent after recanalization
Late MLD change | 3 months
  Changes in mean lumen diameter of the treated vessel, measured up to 5 mm distal to the stent after recanalization and at 3 months follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No
We have planned to perform additional research on this topic.